CLINICAL TRIAL: NCT05588713
Title: A Systematic Study of ADHD Assessments Within Child and Adolescent Psychiatric Care
Brief Title: A Systematic Study of Assessment of Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 467830400
Record Dates: First submitted 2022-09-28; First posted 2022-10-20 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Assessment; Biomarkers; Patient satisfaction; Validity; Reliability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Group A will receive a brief assessment protocol and Group B will receive a comprehensive assessment protocol.
Masking Description: Masking is not possible. The assessors that will review the material for reliability and validity purposes will be blind to diagnostic status of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief assessment protocol (Other): The brief protocol will contain a minimum according to guidelines for assessing ADHD:
  review of medical records, a validated diagnostic interview (MINI-KID), a structured medical history, a pedagogical statement including suspicion of intellectual disability, and rating scales for symptoms such as ADHD, oppositional defiant disorder, autism, anxiety, and depression directed to children (≥ 13 years), parents, and teachers.
  Interventions: Procedure: Brief assessment protocol
- Comprehensive assessment protocol (Other): The comprehensive protocol will extend the brief protocol by adding an approximately three-hour long battery of neuropsychological tests (WISC-V and CPT 3) and biomarkers (heart-rate variability, pupil dilation and the pupillary light reflex) assessed during the CPT 3.
  Interventions: Procedure: Comprehensive assessment protocol

INTERVENTIONS:
Procedure: Brief assessment protocol — The intervention constitutes of a brief assessment protocol for assessing ADHD.
  Arms: Brief assessment protocol
Procedure: Comprehensive assessment protocol — The intervention constitutes of a comprehensive assessment protocol for assessing ADHD.
  Arms: Comprehensive assessment protocol

SUMMARY:
ADHD is one of the most prevalent psychiatric conditions, consuming a large proportion of resources in psychiatric care, often accompanied by long waiting lists to receive proper assessment. The number of ADHD cases has increased, possible due to heightened awareness of the condition. There are large prevalence differences, potentially due to variations in assessments procedures. Many clinicians and parents view the diagnostic process as too extensive, taking time from treatment and interventions. In addition, assessments may be perceived as too focused on diagnostic criteria to be fully helpful. Systematic research on how assessment procedures can be optimized is essentially lacking. It is largely unknown whether brief protocols including medical history, diagnostic interview, and rating scales differ from comprehensive protocols that also encompass neuropsychological testing regarding validity, reliability, patient satisfaction and cost-effectiveness. Further, feasible biomarkers (e.g. heart rate variability, pupil dilation and the pupillary light reflex) of the autonomic nervous system have been proposed as indicators of diagnostic status. The aim of this study is to gain knowledge about diagnostic processes to enable valid, reliable, and cost-effective ADHD assessments. Using a randomized controlled trial design (N = 240 children, 8-17 years, referred to child and adolescent psychiatric units), differences between a brief and a comprehensive ADHD assessment protocol regarding assessment outcome, reliability, validity, patient satisfaction, and future outcome taking gender into account will be examined. The investigators will explore diagnostic sensitivity and specificity of the included assessment instruments and estimate cost-effectiveness of the brief and comprehensive protocols to enable policy makers to make informed decisions. The project will provide important knowledge for patients and clinicians, and inform our understanding of mechanisms underpinning ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years
* Referral for ADHD assessment

Exclusion Criteria:

* Suspected intellectual disability
* Substance abuse
* Psychosis
* Severe depression
* Parent not fluent in Swedish
* Child not living with legal guardian
* Child having protected identity

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Difference in assessment duration between the two protocols | Immediately after completion of assessment
  Numbers of initiated hours to complete the assessments
Difference in prevalence of assigned diagnoses between the two protocols | Immediately after completion of assessment
  Proportion of ADHD diagnoses (including presentation) and comorbid diagnoses
Difference in assessor certainty between the two protocols | Immediately after completion of assessment
  The certainty score will be assigned by the assessor on a 1 to 10-point scale, where 6 to 10 index the assessor's degree of certainty of the child meeting criteria for ADHD and 1 to 5 the assessor's certainty of the child not meeting criteria for ADHD
Difference in reliability between the two protocols | Immediately after completion of assessment
  A second assessor will review the assessment material (blind to diagnostic status) and assign diagnostic status to each case. S/he will be given all information included in the assessment, except for diagnostic status and asked to assign diagnosis/es as well as a certainty score on a 1 to 10-point scale, where 6 to 10 index the assessor's degree of certainty of the child meeting criteria for ADHD and 1 to 5 the assessor's certainty of the child not meeting criteria for ADHD.
Difference in validity between the two protocols | 1 year after completion of assessment
  An experienced clinician will assign diagnostic status using Longitudinal Expert All Data (LEAD; i.e. review of all available material) roughly one year post assessment, after follow-up data has been collected. For this purpose, all available material will include information included in the assessment, medical records following the assessment, and symptom ratings at follow up. S/he will assign diagnosis/es and a certainty score (on a 1 to 10-point scale, where 6 to 10 index the assessor's degree of certainty of the child meeting criteria for ADHD and 1 to 5 the assessor's certainty of the child not meeting criteria for ADHD), blind to original diagnostic status.
Difference in patient satisfaction between the two protocols | Immediately after completion of assessment
  Children (> 13 years) and all legal guardians will rate satisfaction with the assessment process right after the assessment, using a satisfaction scale ranging from 1 to 5, where 5 indicates high satisfaction with the assessment.
Difference in patient satisfaction between the two protocols at follow-up | 1 year after completion of assessment
  Children (> 13 years) and all legal guardians will rate satisfaction with the assessment process at follow up, using a satisfaction scale ranging from 1 to 5, where 5 indicates high satisfaction with the assessment.
Difference in cost effectiveness between the two protocols | 1 year after completion of assessment
  To enable cost-effectiveness analyses, a health economist will build a model based on the following: Child (> 13 years) and parent ratings of child quality of life at baseline and follow-up using the Child Health Utility D9 (CHUD-9), on a scale from 1 to 5, where 1 indicates high quality of life. CHUD-9 will be used to estimate quality adjusted life years (QALYs). Personnel resources and overheads will be estimated for each protocol, and other inputs (such as risks of negative school outcomes and related costs, as well as costs related to ADHD treatment) will be collected from the literature. Consumption of healthcare and school resources for children, as well as productivity losses associated with absenteeism and presentism at school will be estimated from the Treatment Inventory of Costs in Patients (TIC-P), which will be filled out by the caregivers and teachers.

SECONDARY OUTCOMES:
Sensitivity and specificity of the diagnostic interview in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for the diagnostic interview, Mini Internationell Neuropsykiatrisk Intervju (MINI-kid), using formal diagnosis as the external criterion.
Sensitivity and specificity of the ADHD-symptom rating scale in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for the Adult ADHD Self-Report Scale Adolescent version (ASRS-A), in which symptoms are rated on a scale from 1-5, where 5 indicate high symptoms, with formal diagnosis as the external criterion.
Sensitivity and specificity of workning memory in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for the working memory index from Wechlser Intelligence Scale for Children (WISC-V), on a scale from 1 to 19, where 19 indicated high ability for workning memory. Formal diagnosis will be used as the external criterion.
Sensitivity and specificity of Continous Performance Test in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for the Conners Continous Performance Test (CPT-3). The CPT-3 renders a T-score ranging from 0-100, where 50 is the mean and 15 the standard diviation. Higher scores indicate better attention abilities. Formal diagnosis will be used as the external criterion.
Sensitivity and specificity of heart rate variability in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for heart rate variability assessed during the Conners Continous Performance Test (CPT-3). Formal diagnosis will be used as the external criterion.
Sensitivity and specificity of pupil dilation in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for pupil dilation assessed with an eye-tracker during the Conners Continous Performance Test (CPT-3). Formal diagnosis will be used as the external criterion.
Sensitivity and specificity of the pupillary light reflex in relation to ADHD diagnosis | At baseline
  Discriminative validity (positive predictive value, sensitivity, specificity, and area under the curve) will be calculated for the pupillary light reflex. Formal diagnosis will be used as the external criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Matilda Frick, PhD, Principal Investigator — Uppsala University
Locations (1):
- Child and adolescent psychiatry unit, Uppsala, Sweden